CLINICAL TRIAL: NCT03536858
Title: Social Networks and Renal Education: Promoting Transplantation
Acronym: SNARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 11648
Record Dates: First submitted 2018-05-02; First posted 2018-05-25 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: End Stage Renal Disease; Living Donor Kidney Transplantation; Renal Dialysis
Keywords: End Stage Renal Disease; Hemodialysis; Social Network
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Transplantation

STUDY DESIGN:
Intervention Model Description: The investigators will assign every HD clinic shift to one of the two targeting strategies. They will measure the spread of information, attitudes, and behaviors by comparing the patients targeted to participate in the living donor intervention to the other patients on their shift.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Hemodialysis staff will be unaware as to whether the patient was targeted based on their network centrality or clustering. Survey administrators will be unaware of which patient received the living donor intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centrality (Active Comparator): The patients at clinic one who receive hemodialysis on Tuesday, Thursday, Saturday and the patients on the Monday, Wednesday, Friday schedule at clinic two, will be assigned to the Centrality arm. Two patients per hemodialysis shift with the highest centrality will be selected to participate in the COACH (Communicating about Choices in Transplantation) intervention. The patients selected by centrality will have a centrality greater than 1 standard deviation (SD) from the mean of the other patients on their hemodialysis clinic shift and a clustering less than 1 SD from the mean. The investigators will measure the spread of information, attitudes, and behaviors by comparing the targeted patients to the other patients on their shift.
  Interventions: Behavioral: COACH (Communicating about Choices in Transplantation)
- Clustering (Active Comparator): The patients at clinic one who receive hemodialysis on Monday, Wednesday, Friday and the patients on the Tuesday, Thursday, Saturday schedule at clinic two, will be assigned to the Clustering arm.Two patients per hemodialysis shift with the highest clustering coefficient will be selected to participate in the COACH (Communicating about Choices in Transplantation) intervention. The patient selected by clustering coefficient, will have a clustering coefficient greater than 1 SD from the mean of the other patients on their hemodialysis clinic shift and centrality 1 SD less than a mean. The investigators will measure the spread of information, attitudes, and behaviors by comparing the targeted patients to the other patients on their shift.
  Interventions: Behavioral: COACH (Communicating about Choices in Transplantation)

INTERVENTIONS:
Behavioral: COACH (Communicating about Choices in Transplantation) — COACH is a behavioral communication intervention designed specifically for ESRD patients pursuing kidney transplantation. The COACH program consists of four modules: 1) Kidney transplant options, 2) Discussing your transplant options, 3) Requesting living donation, and 4) Maintaining positive relationships. The content and teaching strategies were guided by the concepts of social cognitive theory as well as principles of adult learning and communication skill acquisition. We believe that patients will transfer these skills to other patients at the hemodialysis clinic who are on their shift.

SUMMARY:
There are significant and persistent disparities in access to kidney transplantation and as a result most patients with end stage renal disease receive hemodialysis (HD). HD is unique as it is a treatment performed in a group setting which lends itself to forming social networks. The goal of this research study is to identify and characterize the social networks of HD patients and measure the influence of HD social networks on knowledge, attitudes, and behaviors towards transplantation using repeated surveys and a network targeted educational intervention.

DETAILED DESCRIPTION:
Kidney transplantation is the treatment of choice for end stage renal disease (ESRD). Unfortunately, there are significant and persistent gender and racial disparities in access to transplantation and the successful navigation of transplant evaluation process. The process includes understanding suitability/eligibility for transplantation, obtaining a referral to a transplant center for medical evaluation, completion of medical testing for transplant candidacy, and asking family and friends to donate. Women and ethnic minorities are less likely to be informed of the option of transplantation, referred to a transplant center, and complete the medical evaluation needed to be placed on the kidney transplant waiting list. Modifiable barriers to completing these steps include: lack of knowledge, lack of social support, and inability to discuss transplantation and living donation. As a result chronic hemodialysis (HD) becomes the default treatment. HD clinics are unique social environments in that patients receive their treatments in a group setting which facilitates social networks and the formation of unique micro-communities based on their assigned shift. The robust influences of social networks are well-described in other chronic conditions like obesity, diabetes, and smoking, however, there is scant information on the impact of social networks in HD clinics. Differences in social network structure by gender and race may create critical barriers in the kidney transplant process. White men tend to have diffuse networks which are better for communicating novel information. Women and minorities tend to have clustered/dense networks, which tend to reinforce attitudes and behaviors. It has been speculated that social networks negatively affect transplantation through the clustering of inaccurate information, negative attitudes, and exposure to failed transplants. Our previous observational research, however, suggests that HD patient social network structure can facilitate the completion of pre-transplant steps by providing patients with needed information and support. Further insight into HD social networks has the potential to guide measures to reduce transplant disparities. Our overarching hypothesis is that hemodialysis social networks facilitate the spread of information and behaviors, and that using a targeted social network intervention will improve access to transplantation especially among women and minorities. To address this hypothesis, we will pursue the following specific aims:

Aim 1: Characterize hemodialysis patient social networks by gender and race. Using our previously validated survey, we will model social networks of hemodialysis patients in two independent clinics.

Hypothesis 1: Female hemodialysis patients of all race and ethnicity have dense (higher clustering coefficient) social networks when compared to male HD patients.

Aim 2: Assess the relationship between network structure and knowledge, attitudes, and behaviors towards kidney transplantation. Using the network information from Aim 1, we will analyze the clustering of information, attitudes, and behaviors towards kidney transplantation.

Hypothesis 2: Patients in dense HD clinic social networks have similar attitudes (both positive and negative) about transplantation and behaviors (initiating transplant discussion and completing steps in the kidney transplant process) as compared to patients in diffuse networks.

Aim 3: Compare and contrast the diffusion of knowledge, attitudes, and behaviors regarding transplantation through HD social networks by targeting either the most clustered (as measured by clustering coefficient) or the most central members (as measured by betweenness centrality) of the network to disseminate a transplant education intervention. We will assign every HD clinic shift to one of the two targeting strategies and we will measure the spread of information, attitudes, and behaviors by comparing the targeted patients to the other patients on their shift.

Hypothesis 3: Targeting patients with high clustering coefficient will be the most effective method to spread information and favorable attitudes toward transplantation, as well as completion of steps toward transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older, able to consent to participation and respond to the validated survey in English, and who are present in the HD clinics during the initial survey periods, July 2018 to June 2022 are eligible to participate in the baseline network survey.
* Transplant eligible patients will be eligible to participate. All patients who participate will be evaluated via chart review by a study transplant nephrologist for transplant candidacy and, if eligible, the primary nephrologist will be asked whether the patient is an appropriate candidate and reasons they have not been referred. We will defer the transplant referral to the attending nephrologist. Our criteria for transplant ineligibility are nursing home resident, >79 years of age, active or recent malignancy, inoperable coronary artery disease, or comorbid illness that will make it unlikely that the patient will survive >3 years after transplant.

Exclusion Criteria:

* Patients who are unable or unwilling to provide consent or complete the survey in English .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Primary Knowledge Outcome: Differences in patient knowledge 3 months post-intervention | Baseline to 3 months post intervention
  The investigators will compare the differences in patient transplant knowledge three months post intervention to baseline knowledge. The investigators will compare survey questionnaire answers collected three months post-intervention to those collected pre-intervention. The investigators will use twelve true/false items on transplant knowledge items, summing the correctly answered items to create a composite knowledge score. The higher the composite score the greater the knowledge.
Primary Knowledge Outcome: Differences in patient knowledge 1 year post-intervention | Baseline to 1 year post intervention
  The investigators will compare the differences in patient knowledge regarding transplant one year post intervention to baseline knowledge. The investigators will compare survey questionnaire answers collected one year post-intervention to those collected pre-intervention. They investigators will use twelve true/false items on transplant knowledge items summing the correctly answered items to create a composite knowledge score. The higher the composite score the greater the knowledge.
Primary Behavioral Outcome: Differences in transplant steps completed 3 months post-intervention | Baseline to 3 months post intervention
  The investigators will measure the number of transplant steps completed. The investigators will measure the difference in the transplant step at three months and one year post intervention and compare that to the step prior to the intervention. The steps towards transplant include: 1) transplant suitability for referral to transplant center, 2) interest in transplantation, 3) referral call to transplant center, 4) first visit to transplant center, 5) transplant center work-up, 6) work-up complete, 7) active on the list, 8) successfully received a kidney transplant. A larger number indicates more steps completed.
Primary Behavioral Outcome: Differences in transplant steps completed 1 year post-intervention | Baseline to 1 year post intervention
  The investigators will measure the number of transplant steps completed. The investigators will measure the difference in the transplant step at three months and one year post intervention and compare that to the step prior to the intervention. The steps towards transplant include: 1) transplant suitability for referral to transplant center, 2) interest in transplantation, 3) referral call to transplant center, 4) first visit to transplant center, 5) transplant center work-up, 6) work-up complete, 7) active on the list, 8) successfully received a kidney transplant. A larger number indicates more steps completed.

SECONDARY OUTCOMES:
Completion of transplant work-up 3 months post intervention | 3 months post intervention
  The investigators will confirm with the hemodialysis clinic and the transplant center whether the patient has successfully completed the kidney transplant work-up. This is a binary outcome and will be measured three months.
Completion of transplant work-up 1 year post intervention | 1 year post intervention
  The investigators will confirm with the hemodialysis clinic and the transplant center whether the patient has successfully completed the kidney transplant work-up. This is a binary outcome one year post intervention.
Asking for a living donor 3 months post-intervention | 3 months post intervention
  The investigators will measure patient self-reported requests for living donation, including the number of requests. This will be measured by survey questionnaire three months post intervention
Asking for a living donor 1 year post-intervention | 1 year post intervention
  The investigators will measure patient self-reported requests for living donation, including the number of requests. This will be measured by survey questionnaire one year post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Avrum Gillespie, Principal Investigator — Temple University Hospital
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the final analysis is completed. De-identified data will be available on request from the investigator once proper institutional review board application has been confirmed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 7/2023
Access Criteria: Proposal from researcher

REFERENCES:
- [Background] Gillespie A, Fink EL, Traino HM, Uversky A, Bass SB, Greener J, Hunt J, Browne T, Hammer H, Reese PP, Obradovic Z. Hemodialysis Clinic Social Networks, Sex Differences, and Renal Transplantation. Am J Transplant. 2017 Sep;17(9):2400-2409. doi: 10.1111/ajt.14273. Epub 2017 Apr 21. PMID 28316126
- [Background] Traino HM, West SM, Nonterah CW, Russell J, Yuen E. Communicating About Choices in Transplantation (COACH). Prog Transplant. 2017 Mar;27(1):31-38. doi: 10.1177/1526924816679844. Epub 2016 Nov 25. PMID 27888276
- [Derived] Calvelli H, Gardiner H, Gadegbeku C, Reese P, Obradovic Z, Fink E, Gillespie A. A Social Network Analysis of Hemodialysis Clinics: Attitudes Toward Living Donor Kidney Transplant among Influential Patients. Kidney360. 2024 Apr 1;5(4):577-588. doi: 10.34067/KID.0000000000000383. Epub 2024 Feb 7. PMID 38324254

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03536858/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03536858/SAP_001.pdf